CLINICAL TRIAL: NCT03166865
Title: Clinical Study of Umbilical Cord Mesenchymal Stem Cells (UC-MSC) for Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liaocheng People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: lcsrmyygk
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis (OA); mesenchymal stem cells(MSC)
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intraarticular injection of 2×10~7 Umbilical-cord mesenchimal stem cells with plateler Rich Plasma(5ml)
  Interventions: Biological: Umbilical-cord mesenchymal stromal cells (UC-MSCs)
- Control group (Other): Intraarticular injection of hyaluronic acid
  Interventions: Other: Hyaluronic acid

INTERVENTIONS:
Biological: Umbilical-cord mesenchymal stromal cells (UC-MSCs) — Allogeneic UC-MSCs 1 x 10~7 diluted on 5 mL of Platelet Rich Plasma
  Arms: Intervention group
Other: Hyaluronic acid — intra-articular injection of Hyaluronic Acid
  Arms: Control group

SUMMARY:
Osteoarthritis (OA) is one of the most common joint diseases that is considered a chronic degenerative disorder. There is no effective therapy available today. This prospective clinical trial is designed in an attempt to study the efficacy of mesenchymal stem cells with platelet rich plasma in knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* 30-70 years old.
* No serious infection, chronic diseases, diabetes and tuberculosis.
* Osteoarthritis of the knee with grade1-3 defined by the modified Kellgren-Lawrence classification.
* Written informed consents were obtained from all subjects.

Exclusion Criteria:

* Pregnant women or cognitively impaired adults.
* Inflammatory or post infectious arthritis.
* Intra-articular drug injection within the previous 2 months.
* Serious medical illness with a life expectancy of less than 1 year.
* Prior admission for substance abuse.
* Arthroscopy during the previous 6 months.
* Systemic autoimmune rheumatic disease.
* Poorly controlled diabetes mellitus.
* Immunosuppressive or anticoagulant treatments.
* Treatment with corticosteroids in the 3 months prior to inclusion in the study.
* NSAID therapy within 15 days prior to inclusion in the study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in visual analogue scale (VAS) | Baseline, 1, 3, 6 and 12 weeks
  Visual analogue scale (VAS)
Change From Baseline in western Ontario and McMaster Universities Osteoarthritis Index score | Baseline, 1, 3, 6 and 12 weeks
  WOMAC
Change From Baseline in knee society score (KSS) | Baseline, 1, 3, 6 and 12 weeks
  knee society score (KSS)
Change From Baseline in MOS item short from health survey(SF-36) | Baseline, 1, 3, 6 and 12 weeks
  The MOS item short from health survey(SF-36)

SECONDARY OUTCOMES:
The number of cartilage defects, thickness of cartilage evaluated by X-ray and MRI | Baseline, 1, 3, 6 and 12 weeks
The IL-1β, IL-6, PGE-2, TGF-β, TNF-α and IGF-1 of articular cavity fluid | Baseline, 1, 3, 6 and 12 weeks
  The IL-1β, IL-6, PGE-2, TGF-β, TNF-α and IGF-1 of articular cavity fluid

CONTACTS AND LOCATIONS:
Overall Officials: Dawang Wang, Ph.D., Study Director — Liaocheng People's Hospital
Locations (1):
- Liaocheng city people's hospital, Liaocheng, Shandong, China